CLINICAL TRIAL: NCT06484153
Title: A Randomized Phase 1b/2 Clinical Trial Evaluating Fruquintinib and Pirfenidone in Combination With Anti-PD-1 Antibody in Patients With Standard Treatment Failure of Advanced or Metastatic pMMR/MSS Colorectal Carcinoma
Brief Title: Fruquintinib and Pirfenidone in Combination With Anti-PD-1 Antibody in Advanced or Metastatic pMMR/MSS Colorectal Carcinoma
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Tao Zhang, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: union-P
Record Dates: First submitted 2024-05-24; First posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: To Evaluate the Efficacy of Fruquintinib and Pirfenidone in Combination With Anti-PD-1 Antibody in Colorectal Carcinoma; To Evaluate Whether Pirfenidone Can Reshape the Tumor Microenvironment in Colorectal Cancer; Combination of Fruquintinib and Anti-PD-1 Antibody Was Reported to Improve Patient Prognosis in Colorectal Cancer
Keywords: Pirfenidone,tumor microenvironment, PD-1 antibody
MeSH Terms: interventions — pirfenidone; HMPL-013; pembrolizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Pembrolizumab intravenous (IV) 200mg flat dose day 1 then every 3 weeks. Fruquintinib orally (PO) 3mg po qd.
  Pirfenidone (Esbriet) orally (PO) with food according to this schedule:
  two dose groups: 200mg, TID, po;500mg, TID ,po. Using "3-3" design, the observation period of DLT was 28 days.
  Interventions: Drug: Pirfenidone; Drug: Fruquintinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pirfenidone — Two doses of pirfenidone (200 mg,tid,po;500 mg,tid,po) were set up. Using the 3+3 design, the DLT observation period is 28 days.
Drug: Fruquintinib — 3mg, orally, qd
Drug: Pembrolizumab — 200mg iv every 3 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of fruquintinib and pirfenidone in combination with anti-PD-1 antibody in patients with standard treatment failure of advanced or metastatic pMMR/MSS colorectal adenocarcinoma.

DETAILED DESCRIPTION:
In this study, we explored the potential effectiveness of fruquintinib and pirfenidone in combination with anti-PD-1 antibody, in MSS/pMMR unresectable locally advanced or metastatic colorectal cancer patients who failed standard chemotherapy and testified this new combination in preclinical models. 25 patients were included.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of unresectable locally advanced, recurrent or metastatic colorectal adenocarcinoma.
2. Tumor tissues were identified as mismatch repair-proficient (pMMR) by immunohistochemistry (IHC) method or microsatellite stability (MSS) by polymerase chain reaction (PCR).
3. Subjects must have failed at least two lines of prior treatment.
4. Subjects must have one measurable lesion according to RECIST v1.1 at least.
5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1. 6. 18-75 years old.

7. Life expectancy of at least 12 weeks. 8. Adequate bone marrow, liver, renal and coagulation function as assessed by the laboratory required by protocol

Exclusion Criteria:

1. Previously received anti-programmed death-1 (PD-1) or its ligand (PD-L1) antibody or Pirfenidone.
2. Received last dose of anti-tumor therapy (chemotherapy, targeted therapy, tumor immunotherapy or arterial embolization) within 3 weeks of the first dose of study medication.
3. Received radiotherapy with 4 weeks of the first dose of study medication.
4. Underwent major operation within 4 weeks of the first dose of study medication or open wound, ulcer or fracture.
5. Known symptomatic central nervous system (CNS) metastasis and/or carcinomatous meningitis. Subjects received prior treatment and have stable disease more than 4 weeks from first dose of study medication are permitted to enroll.
6. Active, known or suspected autoimmune disease or has a history of the disease within the last 2 years.
7. Interstitial lung disease requiring corticosteroids.
8. Active or poorly controlled serious infections.
9. Significant malnutrition.
10. Symptomatic congestive heart failure (NYHA Class II-IV) or symptomatic or poorly controlled arrhythmia.
11. Uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 100 mmHg) despite standard treatment.
12. Within 6 months prior to the enrollment, history of gastrointestinal perforation and/or fistula, gastrointestinal ulcer, bowel obstruction, extensive bowel resection, Crohn's disease, or ulcerative colitis, intra-abdominal abscesses, or long-term chronic diarrhea.
13. History or evidence of inherited bleeding diathesis or coagulopathy or thrombus
14. Any life-threatening bleeding within 3 months prior to the enrollment.
15. High risk of bleeding.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-07-22 (Estimated); Primary Completion 2026-07-22 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 year
  The time from enrollment until tumor progression or death from any cause, whichever occurred first
Occurrence of Grade 4 toxicity | Cycle 1 day 1 to Cycle 3 day 1 (Each cycle is 21 days)
  CTCAE v5.0
Occurrence of Grade 3 toxicity | Cycle 1 day 1 to Cycle 3 day 1 (Each cycle is 21 days
  CTCAE v5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | 2 year
  The proportion of patients with a PR or CR
Overall Survival (OS) | 2 year
  The time calculated from enrollment until death from any cause, with living patients censored at the last known survival date
Disease control rate (DCR) | 2 year
  The proportion of patients with a PR, CR, or SD
Duration of response (DoR) | 2 year
  For patients who achieved a complete response (CR) or partial response (PR), the time from the first tumor assessment demonstrating response until disease progression or death, whichever occurred first

IPD SHARING:
Plan to Share IPD: Yes
First use of pirfenidone to unlock the immunosuppressive microenvironment and thereby enhance immunotherapy efficacy in pMMR/MSS colorectal cancer
Supporting Information: Study Protocol
Time Frame: 5 years